CLINICAL TRIAL: NCT04301739
Title: A Randomized, Double-Blind, International Multi-Centre, Phase III Clinical Study to Evaluate Efficacy and Safety of HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) in Combination With Chemotherapy Versus Placebo in Combination With Chemotherapy as Neoadjuvant Therapy and HLX10 Versus Placebo as Adjuvant Therapy in Patients With Triple Negative Breast Cancer (TNBC)
Brief Title: to Evaluate Efficacy and Safety of HLX10 in Combination With Chemotherapy Versus Placebo in Combination With Chemotherapy as Neoadjuvant Therapy and HLX10 Versus Placebo as Adjuvant Therapy in Patients With Triple Negative Breast Cancer (TNBC)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-013-TNBCneo
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Previously Untreated; Potentially Resectable; Without Distant Metastasis
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Doxorubicin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX10 + chemotherapy→ HLX10 (Experimental): HLX10 + chemotherapy (nab-paclitaxel carboplatin) (4 cycles) → HLX10 + chemotherapy (doxorubicin or epirubicin cyclophosphamide) (4 cycles) → surgery → HLX10 (9 cycles)
  Interventions: Drug: HLX10; Drug: nab-paclitaxel, carboplatin, doxorubicin or epirubicin and cyclophosphamide
- Placebo + chemotherapy→ Placebo (Placebo Comparator): Placebo + chemotherapy (nab-paclitaxel carboplatin) (4 cycles) → Placebo + chemotherapy (doxorubicin or epirubicin cyclophosphamide) (4 cycles) → surgery → Placebo (9 cycles)
  Interventions: Drug: nab-paclitaxel, carboplatin, doxorubicin or epirubicin and cyclophosphamide; Drug: Placebo

INTERVENTIONS:
Drug: HLX10 — HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  Arms: HLX10 + chemotherapy→ HLX10
Drug: nab-paclitaxel, carboplatin, doxorubicin or epirubicin and cyclophosphamide — chemotherapeutics
Drug: Placebo — Placebo
  Arms: Placebo + chemotherapy→ Placebo

SUMMARY:
This study is a randomized, double-Blind,international multi-Centre, phase III clinical study to evaluate efficacy and safety of HLX10 in combination with chemotherapy versus placebo in combination with chemotherapy as neoadjuvant therapy and HLX10 versus placebo as adjuvant therapy in previously untreated and potentially resectable patients with TNBC and without distant metastasis.

Eligible subjects in this study will be randomized to Arm A or Arm B at 2:1 ratio as follows:

Arm A (HLX10 arm): HLX10 + chemotherapy (nab-paclitaxel carboplatin) (4 cycles) → HLX10 + chemotherapy (doxorubicin or epirubicin cyclophosphamide) (4 cycles) → surgery → HLX10 (9 cycles) Arm B (placebo arm): Placebo + chemotherapy (nab-paclitaxel carboplatin) (4 cycles) → Placebo + chemotherapy (doxorubicin or epirubicin cyclophosphamide) (4 cycles) → surgery → Placebo (9 cycles) The three stratification factors for randomization include: lymph node metastasis (yes or no), size of primary tumor lesion (T1/T2 or T3/T4), asian population (yes or no).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects histologically diagnosed with previously untreated TNBC (lack of human epidermal growth factor receptor-2 [HER2], estrogen receptor [ER], progesterone receptor expression as determined by the study site).
2. Subjects who are judged as one of the following by the American Joint Committee on Cancer (AJCC) within 4 weeks prior to randomisation:

   1. T1c, N1-N2, M0
   2. T2, N0-N2, M0
   3. T3, N0-N2, M0
   4. T4a-c, N0-N2, M0.
3. Major organs are functioning well
4. Participant must keep contraception

Exclusion Criteria:

1. Subjects with any other active malignancy within 5 years prior to signing the informed consent form or at the same time. Localised tumours that have been cured such as basal cell carcinoma, squamous-cell skin cancer, superficial bladder carcinoma, and cervical cancer in situ are acceptable.
2. Subjects who have received chemotherapy, targeted therapy, or radiotherapy within 12 months prior to the initial dose of the investigational product.
3. Subjects with a history of severe allergy to any monoclonal antibody or investigational product and its excipient.
4. Pregnant or lactating women.
5. Subjects with a known history of psychotropics abuse or drug abuse
6. Subjects presenting other factors not suitable for participation as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2020-04-17 (Estimated); Primary Completion 2022-09-07 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
tumor assessment | up till 5 years after the enroll
  Pathological complete response (pCR) rate (ypT0/Tis, ypN0) (assessed by central pathology laboratory based on American Joint Committee on Cancer (AJCC) staging system)

IPD SHARING:
Plan to Share IPD: No